CLINICAL TRIAL: NCT04566354
Title: Metabolism in Adipose Tissue Followed Following Sprint Exercise
Brief Title: Interleukin-6 Secretion in Adipose Tissue Following Sprint Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Mona Esbjörnsson, Associate Professor, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2015/1054-32
Record Dates: First submitted 2015-09-22; First posted 2020-09-28 (Actual); Last update posted 2020-09-28 (Actual); Status verified 2020-09

CONDITIONS: Metabolism in Adipose Tissue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sprint exercise (Other): Three bouts of 30-s sprint exercise with 20 min rest in between. Three fat biopsies obtained ar rest before first sprint, 15 min after and 120 min after third sprint Blood samples from stomach vein and arteria during the whole experiment
  Interventions: Other: Repeated 30-s sprint exercise

INTERVENTIONS:
Other: Repeated 30-s sprint exercise — Analyze of Interleukin-6 concentration before and after repeated 30-s sprint exercise

SUMMARY:
Low volume sprint exercise training has been shown to reduce body fat despite small total energy expenditure (for ref see Gillen and Gibala 2014). IL-6 has been shown to increase adipose tissue lipolysis in vitro. Therefore, in an initial study on effects of sprint exercise on adipose tissue metabolism the investigators will examine acute short-term exercise effects on adipose tissue IL-6 exchange.

DETAILED DESCRIPTION:
PURPOSE: Low volume sprint exercise training has been shown to reduce body fat despite small total energy expenditure (for ref see Gillen and Gibala 2014). IL-6 has been shown to increase adipose tissue lipolysis in vitro. Therefore, in an initial study on effects of sprint exercise on adipose tissue metabolism the investigators examined acute short-term effects on adipose tissue IL-6 exchange.

METHODS: Four female and four male subjects perform repeated sprint exercise (3 x 30s with 20 min rest between; Wingate-test). Blood samples are repeatedly obtained, up to 120 min after the last sprint (9 min post ex), from catheters inserted percutaneously into brachial artery and a superficial subcutaneous vein on the anterior abdominal wall providing access to the venous drainage from the subcutaneous adipose tissue and analyzed for IL-6 by ELISA and lactate by spectrophotometry. Fat biopsies from the stomach will be obtained before, 15 min and 120 min after the last sprint. Blood flow will be determined by administration of Xenon-133 in the adipose tissue of the stomach. The release rate of Xenon-133 will be registrated continuously during the total investigation.

SUPPORT: This study is supported by grants from the Swedish National Center for Research in Sports

ELIGIBILITY:
Inclusion Criteria:

* Physical active
* Healthy

Exclusion Criteria:

* Smokers
* Pregnant
* On medication
* No infection
* No asthma

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2015-09; Primary Completion 2016-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Il-6 secretion in adipose tissue before and after 30-s repeated sprint exercise | Before 30-s repeated sprint exercise
  Stomach fat biopsies and arterial and stomach vein blood are obtained
Il-6 secretion in adipose tissue before and after 30-s repeated sprint exercise | After 30-s repeated sprint exercise
  Stomach fat biopsies and arterial and stomach vein blood are obtained

SECONDARY OUTCOMES:
Changes in blood flow in adipose tissue | Before 30-s repeated sprint exercise
  Xenon-133 is administered by a subcutaneous injection into the abdominal adipose tissue of approximately 1-2 MBq of Xenon-133 in the form of gas, at rest before work.
Changes in blood flow in adipose tissue | After 30-s repeated sprint exercise
  The rinsing rate of Xenon-133 from the tissue depot is continuously recorded during the study period by a non-invasive method using a portable scintillation detector system (Mediscint) up to 60 minutes after the last sprint work.
Changes in different metabolites | Before 30-s repeated sprint exercise
  Analysed for lactate, ammonia and IL-6
Changes in different metabolites | After 30-s repeated sprint exercise
  Analysed for lactate, ammonia and IL-6

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska Institutet/Karolinska University Hospital, Stockholm, Sweden